CLINICAL TRIAL: NCT04994184
Title: Scoring System in Predicting Perforated Duodenal Ulcer Morbidity and Mortality in Bpkihs
Status: Completed | Type: Observational
Sponsor: B.P. Koirala Institute of Health Sciences (Other)
Responsible Party: Principal Investigator, Nirmal Prasad Sah, Assistant Professor, B.P. Koirala Institute of Health Sciences
Other Study IDs: 2095/020
Record Dates: First submitted 2021-07-29; First posted 2021-08-06 (Actual); Last update posted 2021-08-09 (Actual); Status verified 2021-08

CONDITIONS: Perforated Duodenal Ulcer
Keywords: PULP; Boey; ASA; Perforated duodenal ulcer; Risk score

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Perforated duodenal ulcer: MORBIDITY AND MORTALITY

SUMMARY:
Different scoring systems were developed for risk prediction and adjustment of morbidity from perforated duodenal ulcer. However, these scoring systems are not routinely used in perforated duodenal ulcer patient in everyday clinical practice. Identification of patient with a high risk of adverse outcomes following surgery is important for clinical decision-making which can assist in risk stratification and triage e.g. timing and extent of pre-operative respiratory and circulatory stabilization, postoperative admission to a high dependency unit (HDU), the level and extent of monitoring, and inclusion in specific perioperative care protocols.

Few studies assessed and compared the accuracy indices of PULP with BOEY and ASA in predicting post PPU repair 30-day morbidity Further, the efficacy must be verified in individual settings like ours. So we wish to assess its efficacy in BPKIHS-a tertiary referral center of eastern Nepal.

DETAILED DESCRIPTION:
Perforated peptic ulcer disease (PPU) is an important indication for emergency surgery, complicating 2%-10% of peptic ulcer disease. In the context of modern peptic ulcer therapy, the incidence of PPU has been declining over the past two decades, but mortality has not followed a commensurate decline, in spite of advances in operative strategy and perioperative care.

Omental patch repair of duodenal ulcer perforation is both simpler than and as effective as definitive ulcer surgery in the emergency situation.

However,mortality due to ulcer perforation treated by simple closure and/or other methods is still around 10%. Factors reported to affect mortality in duodenal ulcer perforations in other series are old age, co-morbidity, preoperative hypotension, large size of the perforation, delay in presentation, and, delay in operation .

Several scoring systems have been proposed for the predictions of 30-day morbidity and mortality of perforated peptic ulcer (PPU) in order to risk stratify patients subject to their anticipated complications, and accordingly direct the required attention to high-risk patients. Scoring systems most commonly used include ASA (American Society of Anesthesiologists), Boey and peptic ulcer perforation score (PULP). Each comprises 3-11 demographic, clinical and biochemical variables that consider only pre-operative, or include pre/intra -operative and laboratory findings. Clinical scoring systems need good diagnostic accuracy in order to risk stratify patients correctly.

ELIGIBILITY:
Inclusion Criteria:

* All patient with perforated duodenal ulcer managed surgically

Exclusion Criteria:

* Perforated other organs eg: gastric ulcer or intestinal perforation Incomplete data available in database

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Perforated duodenal ulcer patient who were managed surgically
Sampling Method: Non-Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2021-03-25 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Post PDU repair 30 day morbidity | 30 day
Post PDU repair 30 day mortality | 30 day

CONTACTS AND LOCATIONS:
Locations (1):
- Nirmal Prasad sah, Dharān, Koshi, Nepal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Menekse E, Kocer B, Topcu R, Olmez A, Tez M, Kayaalp C. A practical scoring system to predict mortality in patients with perforated peptic ulcer. World J Emerg Surg. 2015 Feb 21;10:7. doi: 10.1186/s13017-015-0008-7. eCollection 2015. PMID 25722739
- [Result] Moller MH, Engebjerg MC, Adamsen S, Bendix J, Thomsen RW. The Peptic Ulcer Perforation (PULP) score: a predictor of mortality following peptic ulcer perforation. A cohort study. Acta Anaesthesiol Scand. 2012 May;56(5):655-62. doi: 10.1111/j.1399-6576.2011.02609.x. Epub 2011 Dec 23. PMID 22191386
- [Result] Saafan T, El Ansari W, Al-Yahri O, Eleter A, Eljohary H, Alfkey R, Hajjar M, Toffaha A, El Osta A. Assessment of PULP score in predicting 30-day perforated duodenal ulcer morbidity, and comparison of its performance with Boey and ASA, a retrospective study. Ann Med Surg (Lond). 2019 May 10;42:23-28. doi: 10.1016/j.amsu.2019.05.001. eCollection 2019 Jun. PMID 31193430
- [Result] Lohsiriwat V, Prapasrivorakul S, Lohsiriwat D. Perforated peptic ulcer: clinical presentation, surgical outcomes, and the accuracy of the Boey scoring system in predicting postoperative morbidity and mortality. World J Surg. 2009 Jan;33(1):80-5. doi: 10.1007/s00268-008-9796-1. PMID 18958520
- [Result] Makela JT, Kiviniemi H, Ohtonen P, Laitinen SO. Factors that predict morbidity and mortality in patients with perforated peptic ulcers. Eur J Surg. 2002;168(8-9):446-51. doi: 10.1080/110241502321116424. PMID 12549682
- [Result] Kim JM, Jeong SH, Lee YJ, Park ST, Choi SK, Hong SC, Jung EJ, Ju YT, Jeong CY, Ha WS. Analysis of risk factors for postoperative morbidity in perforated peptic ulcer. J Gastric Cancer. 2012 Mar;12(1):26-35. doi: 10.5230/jgc.2012.12.1.26. Epub 2012 Mar 30. PMID 22500261